CLINICAL TRIAL: NCT05729945
Title: Catholic Health Initiatives (CHI) St. Joseph's Children Home Visiting Longitudinal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2250030226
Record Dates: First submitted 2023-01-06; First posted 2023-02-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Child Development; Child Behavior; Child Abuse; Child Neglect; Parenting; Delinquency; Criminal Behavior
Keywords: Home Visiting
MeSH Terms: conditions — Child Behavior; Criminal Behavior | interventions — House Calls

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Visiting Group (Experimental): The home visiting group receives the program interventions which comprises home visits.
  Interventions: Behavioral: home visiting
- Business as Usual Group (No Intervention): The control group is business as usual and does not receive the program intervention.

INTERVENTIONS:
Behavioral: home visiting — The intervention is a three year program that serves families and their first born children through home visiting using paraprofessionals to deliver a hybrid curriculum using the Partners for a Healthy Baby curriculum developed by Florida State University in January 2015.
  Arms: Home Visiting Group

SUMMARY:
This study involves a long-term outcome study of the Catholic Health Initiative St. Joseph's Children (CHI SJC) program using a randomized control study.

The purpose of this study is to determine the short-term and long-term impact and effectiveness of the CHI SJC program. The CHI SJC program has not been studied to determine program effectiveness. The investigators intend to follow families and their children until the children in the study graduate from high-school or turn 19 years of age.

The study, as a template, uses the eight outcome domains listed and described in the Home Visiting Evidence of Effectiveness website (http://homvee.acf.hhs.gov/outcomes.aspx). These eight domains are:

* Child development and school readiness
* Family economic self-sufficiency
* Maternal health
* Reductions in child maltreatment
* Child health
* Linkages and referrals
* Positive parenting practices
* Reductions in juvenile delinquency, family violence, and crime

The investigators expect to observe significant differences among the two groups with respect to the primary outcome domains listed. The investigators expect study group members randomized to the CHI SJC program will perform better on the eight outcome domains.

Other hypotheses include:

Other Hypotheses:

Hypothesis 1. Randomization to CHI SJC will be associated with higher quality functioning and better child health and well-being.

Hypothesis 2. Randomization to CHI SJC will result in more connections to community resources.

Hypothesis 3. Randomization to CHI SJC will result in improved indications of maternal health and positive parenting practices.

Hypothesis 4. Randomization to CHI SJC will be associated with higher measures of family economic self-sufficiency.

Hypothesis 5. Randomization to CHI SJC will be associated with increased school readiness and school progress and attainment.

Hypothesis 6. Randomization to CHI SJC will be associated with reductions in juvenile delinquency, family violence, and crime.

The study will collect outcome data in the same way and, at the same time, from treatment and control group members. Data collection will primarily be comprised of a set of self-report questionnaires and a review of administrative records that target the outcome domains described earlier. Study group members will be assessed at baseline, 6 months, 12 months, 18 months, 24 months, 3 years, 5 years, 8 years, 12 years, 15 years, and at high-school graduation or 19 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Must be first-born child of one of the parents.
* Child must be 3-months of age or less at the time of enrollment.
* At the time of enrollment family must live within the 3 county area covered by the program.

Exclusion Criteria:

* Children older than 3-months.
* Children who are not the first-born child of one of the parents.

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 343 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2038-12-04 (Estimated); Study Completion 2038-12-05 (Estimated)

PRIMARY OUTCOMES:
Child development and school readiness - Child Behavior Checklist (CBCL) to Measure Change at Time Frame Points | 5 years, 8 years, 12 years, 15 years
  The CBCL is widely used to identify problem behavior in children. Problems are identified by a respondent who knows the child well, usually a parent or other caregiver. There are two versions of the checklist. The preschool checklist is intended for use with children aged 18 months to 5 years. The school-age version is for children aged 6 to 18 years. Administration takes 10 to 15 minutes. The checklist uses a 3 point scale (minimum 1 to maximum 3) with higher scores indicating a worse outcome.
  The CBCL is made up of eight syndrome scales:
  * anxious/depressed
  * depressed
  * somatic complaints
  * social problems
  * thought problems
  * attention problems
  * rule-breaking behavior
  * aggressive behavior
  These group into two higher order factors-internalizing and externalizing.
  The 2001 revision added six DSM-oriented scales:
  * affective problems
  * anxiety problems
  * somatic problems
  * ADHD
  * oppositional defiant problems
  * conduct problems
Child Development and School Readiness - Ages and Stages Questionnaire (ASQ) to Measure Change at Time Frame Points | Birth/baseline, 6 months, 12 months, 18 months, 24 months, and 36 months
  The Ages and Stages Questionnaires (ASQ) provide reliable, accurate developmental and social-emotional screening for children between birth and age 6. The ASQ is designed to pinpoint developmental progress and catch delays in young children. The core of the ASQ is 21 questionnaires, each with 30 items that correspond to age intervals from birth to 6 years. The ASQ has been validated in many countries and translated into numerous languages. The ASQ takes between 10 and 15 minutes to administer.
  The parent-completed questionnaires are designed to screen the developmental performance of children in the areas of:
  1. communication,
  2. gross motor skills,
  3. fine motor skills,
  4. problem solving, and
  5. personal-social skills
  The form uses a 3 point scale (minimum 1 to maximum 3) with lower scores indicating a worse outcome.
Child Development and School Readiness - School Records to Measure Change at Time Frame Points | 5 years, 8 years, 12 years, and 15 years
  Review of school records including standardized test scores, and grades. Standardized test scores, and grades will be combined to measure academic growth.
Maternal Health - Edinburgh Postnatal Depression Scale | Baseline/Birth
  Maternal health will be measured using the Edinburgh Postnatal Depression Scale (EDPS). The EDPS is a 10 item questionnaire developed to identify women who may have postpartum depression. A very high EPDS score could suggest a crisis, other mental health issues or unresolved trauma.
  The Edinburgh Postnatal Depression Scale is a widely used screening tool for postpartum depression. The form uses a 3-point scale (minimum 1 to maximum 3) and higher overall scores indicate depression.
Maternal Health - Brief Symptom Inventory | Baseline/Birth
  The Brief Symptom Inventory (BSI), a brief psychological self-report symptom scale and will be used to measure maternal stress. The BSI is a 53-item questionnaire covering nine symptom dimensions of depression:
  1. Somatization
  2. Obsession-compulsion
  3. Interpersonal sensitivity
  4. Depression
  5. Anxiety
  6. Hostility
  7. Phobic anxiety
  8. Paranoid ideation
  9. Psychoticism
  The BSI also includes three global indices of distress:
  1. Global Severity Index,
  2. Positive Symptom Distress Index, and
  3. Positive Symptom Total.
  These measure number and intensity of reported symptoms, as well as the current or past level of symptomology. It can be administered in approximately 4 minutes. The BSI uses a 5-point rating scale (minimum 1 to maximum 5) with higher scores indicating a worse outcome.
Maternal Health - CAGE-AID | Baseline/Birth
  The CAGE-AID is a validated substance abuse screening tool used to screen for alcohol and drug use and will be used to measure primary outcomes surrounding substance abuse. The CAGE-AID consists of 4 questions and takes one minute to administer. One or more positive answers to the CAGE-AID are considered a positive screen.
Maternal Health - Program Administrative Records | Baseline/Birth
  Catholic Health Initiatives St. Joseph's Children (CHI SJC) administrative records for study group members collected by CHI SJC staff members, which include breastfeeding information, parent employment and education, and number of emergency room visits. These measures will be combined to measure maternal health.
Child Health - Program Administrative Records | Baseline/Birth
  Catholic Health Initiatives St. Joseph's Children (CHI SJC) administrative records for study group members collected by CHI SJC staff members, which include breastfeeding information, parent employment and education, and number of emergency room visits. These measures will be combined to measure child health.
Child Health - Adult Adolescent Parenting Inventory (AAPI-2) to Measure Change at Time Frame Points | Birth, 6 months, 12 months, 18 months, 24 months, 36 months, and 5 years
  The AAPI-2 is designed to assess the parenting and child-rearing attitudes of adolescents and adults and measures child health. It is a 40 item inventory with five subscales designed to assess the parenting and child-rearing attitudes of adult and adolescent parent and pre-parent populations. It takes, on average, between 10 and 15 minutes to complete. Scores range from 1-10 with lower scores indicating worse outcomes.
  Responses to the AAPI-2 provide an index of risk in five specific parenting and child-rearing behaviors:
  * Construct A - Expectations of Children
  * Construct B - Empathy Towards Children's Needs
  * Construct C - Use of Corporal Punishment as a Means of Discipline
  * Construct D - Parent-Child Role Responsibilities
  * Construct E - Children's Power and Independence
  Adolescents as young as 13 years old can respond to the AAPI-2. The AAPI-2 is a validated and reliable inventory used to assess parenting attitudes.
Child Health - Modified Checklist for Autism in Toddlers (M-CHAT) to Measure Change at Time Frame Points | 6 months, 18 months, 24 months, and 36 months
  The M-CHAT is designed to screen children aged 16 to 30 months for an autism spectrum disorder (ASD). The 23-item, parent-completed form generally takes 5 to 7 minutes to be completed and a brief time for staff to score. All items are scored as "yes"=1 or "no"=0 with higher scores indicating increased risk.
Child Health - Ages and Stages Questionnaire (ASQ) to Measure Change at Time Frame Points | Birth, 6 months, 12 months, 18 months, 24 months, 36 months
  The Ages and Stages Questionnaires (ASQ) provide reliable, accurate developmental and social-emotional screening for children between birth and age 6. The ASQ is designed to pinpoint developmental progress and catch delays in young children. The core of the ASQ is 21 questionnaires, each with 30 items that correspond to age intervals from birth to 6 years. The ASQ has been validated in many countries and translated into numerous languages. The ASQ takes between 10 and 15 minutes to administer.
  The parent-completed questionnaires are designed to screen the developmental performance of children in the areas of:
  1. communication,
  2. gross motor skills,
  3. fine motor skills,
  4. problem solving, and
  5. personal-social skills
  The form uses a 3 point scale (minimum 1 to maximum 3) with lower scores indicating a worse outcome.
Child Health - Abidin Parenting Stress Index Short Form (PSI-SF) to Measure Change at Time Frame Points | 6 month, 12 month, 18 month, 24 month, 36 month
  Child health will be assessed using the Abidin Parenting Stress Index Short Form (PSI-SF). The instrument is a well-validated 36 item measure of perceived stress in the parenting role with sound test-retest reliability and internal consistency. The PSI/SF yields a Total Stress score from three scales:
  1. Parental Distress,
  2. Parent-Child Dysfunctional Interaction, and
  3. Difficult Child.
  Average time to complete is 10 minutes. Each item is rated on a 5 point scale (minimum 1 to maximum 5) with higher scores indicating more stress.
Child Maltreatment - Conflict Tactics Scale Parent-Child Form (CTS-PC) to Measure Change at Time Frame Points | 6 months, 12 months, 18 months, 24 months, 36 months, 5 years, 8 years, 12 years and 15 years
  The CTS-PC is one of the most widely used instruments for identifying domestic violence and will be used to measure child maltreatment. The CTS-PC is a 35 item tool that is intended to measure psychological and physical maltreatment, and neglect of children by parents as well as non violent modes of discipline. Specifically, it measures if a parent has carried out acts of physical and psychological aggression, regardless of whether or not the child is injured. The assessment tool is a self-report measurement tool. The tool uses an 8-point scale (minimum 0 to maximum 7) with higher scores indicating greater conflict.
Reduction in Child Maltreatment - Parenting Sense of Competence (PSOC) to Measure Change at Time Frame Points | 5 years, 8 years, 12 years and 15 years
  The 17-item PSOC can be used to measure program outcomes, and, in other contexts, to measure a parent's level of perceived competence. It can also be used to measure satisfaction in parenting, and confidence in parenting efficacy individually, or as a combined total measure.
  The PSOC was developed to assess parenting self-esteem using two rationally derived scales, as Efficacy and Satisfaction. The Efficacy factor examines the parents' competence, capability levels, and problem-solving abilities in their parental role; the Satisfaction factor examines the parents' anxiety, motivation and frustration. Average time to complete is less than 5 minutes. Each item is scored on a 6-point scale (minimum 1 to maximum 6) with higher scores equaling greater self-esteem.
Reductions in Child Maltreatment - New Mexico Children, Youth and Families Department records to Measure Change at Time Frame Points | 6 months, 12 months, 18 months, 24 months, 36 months, 5 years, 8 years, 12 years, and 15 years
  New Mexico Children, Youth and Families Department (CYFD) data for any record of services received that include involvement in the Protective Services Division (PSD), early childhood services, or juvenile justice services. This includes abuse and neglect data. These measures will be combined to measure changes in child maltreatment at listed time frames.
Linkages and referrals - NM Human Services Department (HSD) records to Measure Change at Time Frame Points | Birth, 12 months, 18 months, 24 months, and 36 months
  Review of HSD records (i.e., SNAP, housing, medical, GED, etc.). These measures will be combined to measures linkages and referrals to community resources at listed time frames.
Positive parenting practice - Brief Symptom Inventory | Baseline/Birth
  The Brief Symptom Inventory (BSI), a brief psychological self-report symptom scale and will be used to measure maternal stress. The BSI is a 53-item questionnaire covering nine symptom dimensions of depression:
  1. Somatization
  2. Obsession-compulsion
  3. Interpersonal sensitivity
  4. Depression
  5. Anxiety
  6. Hostility
  7. Phobic anxiety
  8. Paranoid ideation
  9. Psychoticism
  The BSI also includes three global indices of distress:
  1. Global Severity Index,
  2. Positive Symptom Distress Index, and
  3. Positive Symptom Total.
  These measure number and intensity of reported symptoms, as well as the current or past level of symptomology. It can be administered in approximately 4 minutes. The BSI uses a 5-point rating scale (minimum 1 to maximum 5) with higher scores indicating a worse outcome.
Positive Parenting Practices - Adult Adolescent Parenting Inventory (AAPI-2) to Measure Change at Time Frame Points | Birth, 6 months, 12 months, 18 months, 24 months, 36 months, and 5 years
  The AAPI-2 is designed to assess the parenting and child-rearing attitudes of adolescents and adults and measures child health. It is a 40 item inventory with five subscales designed to assess the parenting and child-rearing attitudes of adult and adolescent parent and pre-parent populations. It takes, on average, between 10 and 15 minutes to complete. Scores range from 1-10 with lower scores indicating worse outcomes.
  Responses to the AAPI-2 provide an index of risk in five specific parenting and child-rearing behaviors:
  * Construct A - Expectations of Children
  * Construct B - Empathy Towards Children's Needs
  * Construct C - Use of Corporal Punishment as a Means of Discipline
  * Construct D - Parent-Child Role Responsibilities
  * Construct E - Children's Power and Independence
  Adolescents as young as 13 years old can respond to the AAPI-2. The AAPI-2 is a validated and reliable inventory used to assess parenting attitudes.
Family Economic Self-Sufficiency - N.M. Human Services Department (HSD) | Birth, 6 months, 12 months, 24 months, 36 months, 5 years, and 8 years
  Review of HSD records for public assistance (i.e., SNAP, housing, medical, GED, etc.) and program records of care-giver/parent reports of economic measures (i.e., SES, employment, education, use of community services, etc.), and family stability (i.e., relationship length, marital status, etc.).
Reductions in juvenile delinquency, family violence, and crime - Conflict Tactics Scale Parent-Child Form (CTS-PC) | 6 months, 12 months, 24 months, 36 months, 5 years, 8 years, 12 years, and 15 years
  The CTS-PC is one of the most widely used instruments for identifying domestic violence and will be used to measure child maltreatment. The CTS-PC is a 35 item tool that is intended to measure psychological and physical maltreatment, and neglect of children by parents as well as non violent modes of discipline. Specifically, it measures if a parent has carried out acts of physical and psychological aggression, regardless of whether or not the child is injured. The assessment tool is a self-report measurement tool. The tool uses an 8-point scale (minimum 0 to maximum 7) with higher scores indicating greater conflict.
Changes in juvenile delinquency, family violence, and crime - Jail data | 18 years up to 19 years
  Jail data for any booking records that includes the booking date, release date, and booking charges.
Changes in juvenile delinquency, family violence, and crime - Law Enforcement records | 18 years up to 19 years
  Law enforcement data that will include the date of each arrest, whether the individual was transported to Jail or cited/summoned, and the arrest charges.
Changes in juvenile delinquency, family violence, and crime - Court records | 18 years up to 19 years
  Public court records that include the filing of all criminal cases that will include the date of filing, charges, case closing date, and case disposition.
Changes in juvenile delinquency, family violence, and crime - Children, Youth and Families Department (CYFD) data | 8 years up to 18 years
  CYFD data for any record of services received that include involvement in the Protective Services Division (PSD), early childhood services, or juvenile justice services.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Guerin, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No